CLINICAL TRIAL: NCT04563975
Title: Toripalimab Combined With Docetaxel or Nab-paclitaxel in the Treatment of Advanced Gastric Cancer : a Single-arm, Open Label, Prospective Phase II Clinical Trial
Brief Title: Efficacy and Safety of Toripalimab Combined With Docetaxel or Nab-paclitaxel in Patients With Advanced Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tao Zhang (Other)
Responsible Party: Sponsor-Investigator, Tao Zhang, Chief Physician, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Organization: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XHZL-0236-02
Record Dates: First submitted 2020-09-20; First posted 2020-09-25 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Gastric Cancer Stage IV
MeSH Terms: conditions — Stomach Neoplasms | interventions — toripalimab; Docetaxel; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chemotherapy and programmed death 1 inhibitor (Experimental): Docetaxel /nab-paclitaxel in combination with Toripalimabs
  Interventions: Drug: Toripalimab; Drug: Docetaxel; Drug: nab-paclitaxel

INTERVENTIONS:
Drug: Toripalimab — Toripalimab，240mg，d1，Intravenous Infusion，q3w
  Other Names: JS001
Drug: Docetaxel — Docetaxel，60-75mg/m2，d8 and d15，Intravenous Infusion，q3w
  Other Names: Taxotere
Drug: nab-paclitaxel — nab-paclitaxel，125mg/m2，d1 and d 8，Intravenous Infusion，q3w
  Other Names: AI YUE

SUMMARY:
The single arm clinical study is to evaluate the efficacy and safety of an anti-PD-1 antibody (Toripalimab) combined with chemotherapy (docetaxel or nab-Paclitaxel) in patients with advanced gastric cancer who failed first-line treatment.

DETAILED DESCRIPTION:
54 patients who meet the inclusion criteria will receive Docetaxel (60-75mg/m2, every 3 weeks) or nab-Paclitaxel （125mg/m2，every 3 weeks）combined with Toripalimab( 240mg,every 3 weeks）for 4-8 cycles until the disease progresses or intolerable toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18-75
2. Written informed consent from the patient.
3. Pathologically diagnosed gastric or gastroesophageal junction adenocarcinoma (GEJ).
4. Failure of first-line chemotherapy with fluorouracil ，or adjuvant therapy with fluorouracil drugs, but the end of adjuvant treatment is less than 6 months.
5. Measurable disease as per RECIST 1.1 criteria.
6. Adequate organ and bone marrow functions.
7. Female subjects should agree to use a medically approved effective contraceptive during the study period and for up to 6 months after the study，and must undergo a serum-negative pregnancy test within 72hours before starting the study drug, and out of lactation;male subjects should agree to use medically approved methods of contraception during the study period and within 6 months after the end of the study period.
8. Performance Status(ECOG) 0-2.
9. Life expectancy >3 months.

Exclusion Criteria:

1. First-line treatment with Taxanes- containing drugs.
2. Patients with any history of known or suspected autoimmune disease with the specific exceptions of vitiligo, atopic dermatitis, or psoriasis not requiring systemic treatment.
3. Have received immunosuppressive drugs within 2 weeks before starting the study drug, excluding local glucocorticoids or systemic glucocorticoids<10 mg/day prednisone or other glucocorticoids of equivalent dose.
4. Patients with HIV-positive.
5. Patients with viral hepatitis (such as HBV（hepatitis B virus）, HCV（hepatitis C virus）), HBV-DNA> 2000IU/mL, and unwilling to receive antiviral treatment.
6. History of clinically-significant cardiovascular disease ，Liver diseases such as liver cirrhosis decompensated liver disease, and chronic active hepatitis; poorly controlled diabetes (fasting blood glucose (FBG)>10mmol/L); urine routine indicates urine protein ≥++, and 24-hour urine protein quantitative > 1.0g.
7. Clinically-significant pulmonary compromise, including a requirement for supplemental oxygen use to maintain adequate oxygenation.
8. History of (non-infectious) pneumonitis that required steroids or presence of active pneumonitis.
9. History of prior allogeneic bone marrow, stem-cell or solid organ transplantation.
10. Clinically-significant gastrointestinal disorders, such as perforation, gastrointestinal bleeding, or diverticulitis.
11. History of malignant tumors (except for skin basal cell carcinoma and cervical carcinoma in situ treatment with tumor-free survival for more than 3 years.
12. patients with uncontrollable seizures, or loss of insight due to mental illness.
13. History of severe allergies or specific constitution.
14. Participant in other clinical trials within 28 days before study treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2020-07-02 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
disease control rate | At 12 weeks
  disease control rate，According with RECIST 1.1

SECONDARY OUTCOMES:
progression free survival | Up to 12months
  progression free survival
Complication Rate | Up to 12months
  Complication Rate
overall survival rate | one year
  overall survival rate

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Center, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] HAENSZEL W. Variation in incidence of and mortality from stomach cancer, with particular reference to the United States. J Natl Cancer Inst. 1958 Aug;21(2):213-62. No abstract available. PMID 13576088
- [Background] Ter Veer E, Haj Mohammad N, van Valkenhoef G, Ngai LL, Mali RMA, Anderegg MC, van Oijen MGH, van Laarhoven HWM. The Efficacy and Safety of First-line Chemotherapy in Advanced Esophagogastric Cancer: A Network Meta-analysis. J Natl Cancer Inst. 2016 Aug 30;108(10). doi: 10.1093/jnci/djw166. Print 2016 Oct. PMID 27576566
- [Background] Ford HE, Marshall A, Bridgewater JA, Janowitz T, Coxon FY, Wadsley J, Mansoor W, Fyfe D, Madhusudan S, Middleton GW, Swinson D, Falk S, Chau I, Cunningham D, Kareclas P, Cook N, Blazeby JM, Dunn JA; COUGAR-02 Investigators. Docetaxel versus active symptom control for refractory oesophagogastric adenocarcinoma (COUGAR-02): an open-label, phase 3 randomised controlled trial. Lancet Oncol. 2014 Jan;15(1):78-86. doi: 10.1016/S1470-2045(13)70549-7. Epub 2013 Dec 10. PMID 24332238
- [Background] Fuchs CS, Doi T, Jang RW, Muro K, Satoh T, Machado M, Sun W, Jalal SI, Shah MA, Metges JP, Garrido M, Golan T, Mandala M, Wainberg ZA, Catenacci DV, Ohtsu A, Shitara K, Geva R, Bleeker J, Ko AH, Ku G, Philip P, Enzinger PC, Bang YJ, Levitan D, Wang J, Rosales M, Dalal RP, Yoon HH. Safety and Efficacy of Pembrolizumab Monotherapy in Patients With Previously Treated Advanced Gastric and Gastroesophageal Junction Cancer: Phase 2 Clinical KEYNOTE-059 Trial. JAMA Oncol. 2018 May 10;4(5):e180013. doi: 10.1001/jamaoncol.2018.0013. Epub 2018 May 10. PMID 29543932
- [Background] Kato K, Satoh T, Muro K, Yoshikawa T, Tamura T, Hamamoto Y, Chin K, Minashi K, Tsuda M, Yamaguchi K, Machida N, Esaki T, Goto M, Komatsu Y, Nakajima TE, Sugimoto N, Yoshida K, Oki E, Nishina T, Tsuji A, Fujii H, Kunieda K, Saitoh S, Omuro Y, Azuma M, Iwamoto Y, Taku K, Fushida S, Chen LT, Kang YK, Boku N. A subanalysis of Japanese patients in a randomized, double-blind, placebo-controlled, phase 3 trial of nivolumab for patients with advanced gastric or gastro-esophageal junction cancer refractory to, or intolerant of, at least two previous chemotherapy regimens (ONO-4538-12, ATTRACTION-2). Gastric Cancer. 2019 Mar;22(2):344-354. doi: 10.1007/s10120-018-0899-6. Epub 2018 Dec 1. PMID 30506519
- [Background] Langer CJ, Gadgeel SM, Borghaei H, Papadimitrakopoulou VA, Patnaik A, Powell SF, Gentzler RD, Martins RG, Stevenson JP, Jalal SI, Panwalkar A, Yang JC, Gubens M, Sequist LV, Awad MM, Fiore J, Ge Y, Raftopoulos H, Gandhi L; KEYNOTE-021 investigators. Carboplatin and pemetrexed with or without pembrolizumab for advanced, non-squamous non-small-cell lung cancer: a randomised, phase 2 cohort of the open-label KEYNOTE-021 study. Lancet Oncol. 2016 Nov;17(11):1497-1508. doi: 10.1016/S1470-2045(16)30498-3. Epub 2016 Oct 10. PMID 27745820
- [Background] Shitara K, Ozguroglu M, Bang YJ, Di Bartolomeo M, Mandala M, Ryu MH, Fornaro L, Olesinski T, Caglevic C, Chung HC, Muro K, Goekkurt E, Mansoor W, McDermott RS, Shacham-Shmueli E, Chen X, Mayo C, Kang SP, Ohtsu A, Fuchs CS; KEYNOTE-061 investigators. Pembrolizumab versus paclitaxel for previously treated, advanced gastric or gastro-oesophageal junction cancer (KEYNOTE-061): a randomised, open-label, controlled, phase 3 trial. Lancet. 2018 Jul 14;392(10142):123-133. doi: 10.1016/S0140-6736(18)31257-1. Epub 2018 Jun 4. PMID 29880231